CLINICAL TRIAL: NCT02565563
Title: Digitally Recording Heart Rate Variability Via the Patient's Finger: Is There a Difference Between Eye Movements and no Eye Movements During Eye Movement Desensitisation Reprocessing Treatment for Post Traumatic Stress Disorder?
Brief Title: Recording Heart Rate Variability During Eye Movement Desensitisation Reprocessing With or Without Eye Movement
Acronym: EMDR;PTSD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants recruited
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Tayside (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 173479
Record Dates: First submitted 2015-09-21; First posted 2015-10-01 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2015-09

CONDITIONS: Post Traumatic Stress Disorder
Keywords: EMDR; Mechanisms; Eye Movement Desensitisation Reprocessing
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eye Movements (Active Comparator): Eye Movement Desensitisation Reprocessing with eye movements (measuring Heart Rate Variability using HeartMath)
  Interventions: Other: Eye Movement Desensitisation Reprocessing; Device: HeartMath measuring Heart Rate Variability (HRV)
- No Eye Movements (Active Comparator): Eye Movement Desensitisation Reprocessing without eye movements (measuring Heart Rate Variability using HeartMath)
  Interventions: Other: Eye Movement Desensitisation Reprocessing; Device: HeartMath measuring Heart Rate Variability (HRV)

INTERVENTIONS:
Other: Eye Movement Desensitisation Reprocessing — The purpose of this study is not to assess the device itself. The new device will seek to measure heart rate variabilty during the administration of the treatment EMDR. It will measure the patients sympathetic nervous systems (anxiety arousal). Previous reseach studies have used Electrocardiography (ECG) and the purpose of this study is to determine whether or not this device will obtain similar findings as ECG has done.
Device: HeartMath measuring Heart Rate Variability (HRV) — This small device will be attached to the patients finger to allow their heart rate variability to be measured.

SUMMARY:
The purpose of the study is to gain greater insight into Eye Movement Desensitisation Reprocessing (EMDR). EMDR is an NHS recommended treatment, which can significantly reduce trauma symptoms. There is some debate regarding how it actually works, however there is evidence to suggest that the eye movements component helps reduce anxiety and increase relaxation levels. To measure these arousal levels during EMDR previous research has used electrocardiography (ECG) to measure heart rate, which offers insight into the effectiveness of eye movements (EM). All studies to date have used ECG to measure arousal levels which requires technical knowledge to administer and interpret. Furthermore, applying electrodes to a patient experiencing PTSD may heighten anxiety. The present study will use new technology which is a small device that would be gently attached to the end of the patient's index finger. This device is very similar to one that measures oxygen levels in the blood and therefore is a very simple piece of equipment and should cause no discomfort to the patient. The study also requires patient's faces to be video recorded throughout and it will only be their face that is recorded. This is to match the stages of treatment (i.e. when EM starts and stops) to their corresponding arousal level outcome. The new technology will digitally measure the patient's anxious and relaxed arousal levels during EM and no EM treatment sessions. 10 NHS patients would be recruited to receive two treatment sessions; one with EM and one without and then continue with treatment as usual without any of the recording devices. EM and no EM phases occur at least three times within a treatment session and therefore several measurements can be taken and analysed.

DETAILED DESCRIPTION:
DESIGN Each patient will receive an Eye Movement Desensitisation Reprocessing (EMDR) treatment session with eye movements (EM) and an EMDR treatment session without EM. Half will complete the EM session first and the other half will complete the no EM session first. After the first session is complete the patients will cross over to complete the other treatment session, which will be approximately one week later. This is known as a cross over design and allows patients to act as their own control group. Furthermore they will be randomly allocated into which condition they complete first to reduce order effects. During both treatment sessions patients will have their arousal levels digitally measured and face video recorded.

METHODOLOGY Patients who have been referred for trauma will be allocated from the NHS Tayside waiting list. From January 2013 to January 2014 there were approximately 72 patients across Tayside who were treated for Post Traumatic Stress Disorder (PTSD) and/or 'reaction to severe stress, and adjustment disorders'. This was taken from the online patient database (MiDIS), which is mandatory for all clinicians in NHS Tayside to complete.

PROCEDURE NHS Tayside Adult Psychological Therapies Service receives electronic referrals, usually from the GP, stating the reason for referral. The patients' symptoms/diagnoses and CHI number are then documented in a diary waiting to be allocated to the next available appointment. The clinicians will look through the diary, noting the ones who appear to meet the relevant diagnosis/symptoms to ensure that they will be seen by an EMDR qualified clinician if they choose to be seen by psychology at all. Patient's who appear to meet the initial criteria, will be sent a standard protocol appointment letter, stating that they must contact the service within 2 weeks if they still wish to be seen by psychology. Those who choose to be seen will be provided with an initial assessment session, where information is gathered about their presenting problems and history. They will also be asked to complete routine questionnaires. This will be completed by the EMDR qualified clinician, who at the same time will offer them to take part in the study if they believe the patient is suitable for EMDR. If the therapist believes the patient is not suitable for EMDR then as part of standard protocol the assessment will be completed and the patient will be allocated to the next available clinician for treatment. If the patient is suitable then the clinician will explain the parameters of the study which will include, digitally measuring arousal levels and video recording the patient's face during their first two treatment sessions of EMDR therapy with the assessing clinician. Also at their first session the clinician will show the equipment that will be used and provide them with a participant information letter about the study for them to take away and think about. Within the information letter they will be informed that choosing not to take part will not affect their routine care and even if they choose to take part they can drop out at any time and continue with treatment as usual. The chief investigator's contact details will also be provided, should they require further information. At the end of the letter they will be provided with 2 options: 1. I agree to take part in the study. 2. I do not wish to take part in the study. They will need to contact the service within 5 days of their first session to inform us of their decision. This is to allow the equipment to be set up in advance if they agree to take part. Regardless of whether they decide to take part in the study or not, their next session will be within 2 weeks of the initial assessment, which will be with the same clinician if they take part, but may be a different clinician of they do not take part, which is within standard service protocol.

Those who agree to take part in the study will be required to bring their signed consent form (contained within the participant information letter) to their second session or complete another one on the day before engaging within the study. Their second session will either be to complete the assessment process/other formal measures (documented below) or start with EMDR treatment. This will be up to the clinician depending on how much information was gathered in session 1. This is within standard service protocol. Before treatment can begin each patient must complete the formal assessment measures. Only the 2 treatment sessions will use the recording equipment and following this they will continue with treatment without being part of the study. If at any point they decide that they no longer wish to take part, treatment will continue as usual, without the recording devices.

EMDR trained clinicians will administer the EMDR treatment with 3 or 4 patients each. As standard service protocol, patients will receive a minimum of one hour per treatment session and each session will take place in an NHS psychological therapies service building.

Within the treatment sessions patients will be exposed to EMDR with eye movements (Condition 1, C1) and EMDR without eye movements (Condition 2, C2) conducted by the EMDR accredited therapist. Patients will be randomly allocated into either C1 or C2 for his or her first session. Session one and session two will be no more than two weeks apart with each session lasting approximately one hour. At the beginning of each session patients will be required to attach the small infrared transmittance heart rate sensor (HeartMath) to their index finger, which will digitally record their arousal levels and transfer the responses to the laptop. Their face will also be video recorded during the entire session by a small camera on a laptop located approximately three feet across from them. The purpose of this is to be able to match the time of when specific EMDR phases were administrated (the eye movements), to the same time of the patients HRV response. Although faces will be recorded throughout the entire session, only certain stages of the eight stage therapy protocol will be analysed. A five minute adaptation period will be given to all individuals. During both treatment sessions the therapist will use a chosen life event to use within the EMDR protocol. Where possible, the clinician will seek to ensure that each patient will complete the full eight stage protocol as outlined by Shapiro (1989) (Appendix 1). Each individual will also score the vividness scale before and after each condition is completed. A self measure of distress level (known as subjective units of distress [SUD]) are also obtained throughout each session as part of standard EMDR protocol, requiring the patient to rate their level of distress on a scale of 1 to 10.

MEASURES:

Routinely used within the National Health Service (NHS):

1. Beck's Depression Inventory-II (BDI-II) (Beck et al., 1961) will be administered in session 1, to ascertain the participants' mental health and well being. The BDI-II will be used because it is a widely used measure of depression (Beck et al, 1988).
2. The Life Events Checklist (LEC) (Weathers et al., 2013) will be administered in session 1 or 2, but before treatment commences, to determine a specific trauma that patients have been subjected to within their life. The LEC is a measure of exposure to potentially traumatic events, which was developed at the National Centre for Posttraumatic Stress Disorder (PTSD). Once a trauma has been identified this will be the specific trauma that will be used within treatment.
3. Impact of event scale (IES) (Horowitz et al., 1979) will be completed in session 1 or 2, but before treatment begins. It will be administered in conjunction to the LEC, to measure post trauma symptomology, which is one of the most widely used self-report measures.
4. Patients self measure of distress (also known as Subjective Units of Distress [SUDs]) - This will be measured on a scale of 1 to 10 and is part of the eight stage EMDR protocol. This will occur during the 2 treatment sessions.

Measures not routinely used in the NHS service:

1. Dissociative Experiences Scale (DES) (Bernstein & Putnam): this will be administered in session 1, to screen patients who dissociate, since EMDR is found to be ineffective with patients who dissociate as they are unable to attend to the unpleasant thought. Patients scoring 30 and above will be excluded from this study. Although a formal dissociate measure is not routinely use, therapists will often use their clinical judgement to determine if someone is dissociating.
2. Arousal levels - Heart Rate Variability (HRV) will be digitally recorded using an infrared transmittance heart rate sensor (HeartMath) which will be connected to the patient's index finger throughout the entire 2 treatment sessions. The device is very similar to the device that measures oxygen levels in the blood.
3. Facial Behaviour - A laptop camera, located three feet away from the patient, will record the patient's face throughout the entire 2 treatment sessions, so that the time when the different phases of EMDR are administered can be matched to the same time on the patient's arousal level response. In order to accurately match patients' arousal responses to what treatment phase of EMDR was being administered recording must be achieved. Recording facial behaviour may also allow for other observable analysis to be completed.
4. Vividness Scale - Barrowcliff et al. (2004) found eye movements to produce a greater reduction in arousal and vividness for memories associated with fear and anxiety compared with an eye stationary condition using physiological measures of arousal. It has also been found that eye movements resulted in reduced ratings of distress and vividness compared to a no eye movement condition (Kavanagh et al, 2001). Therefore this study will inform the degree of vividness associated with a particular image by asking the patient to hold the image in mind for ten seconds and then indicate on a ten centimetre visual analogue scale the degree to which the image appeared vivid from ''not clear at all'' to ''very clear''. The scale will contain more than two anchors to provide individuals with greater clarity. This is identical to a procedure used in previous studies on vividness (van den Hout et al., 2001). This will be administered during their 2 treatment sessions.

DATA COLLECTION:

Arousal levels and facial video recordings will be collected by the laptop program. The chief investigator will review and analyse the results in order to determine whether eye movements during EMDR treatment significantly improves arousal levels (i.e. is the patient more relaxed) compared to no eye movements during EMDR treatment. Analysis will also include taking time points across each treatment session in order to determine whether or not arousal levels improve over the course of the session (i.e. do patients anxiety levels reduce over the course of the session).

TIME FRAMES:

Identify patients from waiting list by 1st October 2015. Patients to get in touch by beginning of November to commence treatment end of November 2015 and complete by end of February 2016. Analyse the data by the beginning of March 2016 and then commence write up to complete by end of April 2016.

A pilot study using the same technology and similar method as above was completed with 4 Undergraduate students.

ELIGIBILITY:
Inclusion Criteria:

* Patients on the waiting list for psychological treatment who meet criteria for PTSD and/or sub clinical PTSD.
* Patients over the age of 18.
* Patients able to give informed consent
* Single trauma event

Exclusion Criteria:

* Patients in other psychological treatment.
* Patients unable to provide informed consent
* Patients who are actively suicidal
* Patients who score above 30 on the dissociative experiences scale (DES).
* Difficulties with eye sight, where vision cannot be corrected with glasses or lenses (EMDR requires the patient to accurately follow their finger with their eyes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2016-02 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability (HRV) | up to 7 months
  This is the variation in the beat-to-beat interval and measures the sympathetic nervous system (SNS).
  A minimum of 3 arousal level (HRV) measurements will be taken within each treatment session. An average measurement will be calculated for each patient during each condition. Paired sample t-tests will be used to compare heart rate variability (arousal levels) outcomes between eye movements and no eye movements for each patient.
  A repeated measures ANOVA will be used to analyse any differences across each session of eye movements and no eye movements (containing a minimum of 3 phases in each session), to see if there is an improvement in HRV (i.e. a reduction in anxiety arousal and increase in relaxed arousal) over each session.

SECONDARY OUTCOMES:
Subjective Units of Distress (SUDs) | up to 7 months
  Do patients' self rating scores of distress (within EMDR treatment this is known as subjective units of distress [SUDs]) reduce as their anxiety levels reduce and their relaxation levels increase?
  A test of correlation will be conducted to determine the relationship between patients subjective units of distress and HRV.